CLINICAL TRIAL: NCT01747382
Title: Catheter-based Renal Sympathetic Nerve Ablation for Treatment-resistant Hypertension in Patients With Chronic Kidney Disease
Brief Title: Renal Denervation for Treatment of Resistant Hypertension in Patients With Chronic Kidney Disease
Status: No longer available | Type: Expanded Access
Sponsor: Singapore General Hospital (Other)
Collaborators: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: NKFRC/2011/07/26
Record Dates: First submitted 2012-12-09; First posted 2012-12-11 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Hypertension; Chronic Kidney Disease
Keywords: Treatment-resistant Hypertension; Chronic Kidney Disease; Symplicity catheters; Renal denervation
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

INTERVENTIONS:
Procedure: Renal denervation
  Other Names: Symplicity radiofrequency catheter

SUMMARY:
Recent clinical studies have demonstrated that catheter-based renal sympathetic nerve ablation is safe and effective in treating patients with resistant hypertension. However, there is limited data on its safety and efficacy in patients with Chronic Kidney Disease.

The investigators hypothesize that catheter-based renal sympathetic nerve ablation is safe and effective in the treatment of resistant hypertension in patients with Chronic Kidney Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Individual has a systolic blood pressure ≥ 160 mmHg (≥ 150 mmHg for type 2 diabetics).
2. Individual is adhering to a stable drug regimen including 3 or more anti-hypertensive medications, of which one is a diuretic, (with no changes for a minimum of 2 weeks prior to enrollment) and is expected to be maintained for at least 6 months.
3. Individual with stage 3 chronic kidney disease, defined as having an eGFR of 30 - 60 mL/min/1.73m2, using the MDRD calculation.
4. Individual is ≥ 21 and ≤ 65 years of age.
5. Individual agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

1. Individual has renal artery anatomy that is ineligible for treatment including:

   1. Main renal arteries < 4 mm in diameter or < 20 mm in length.
   2. Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which, in the eyes of the operator, would interfere with safe cannulation of the renal artery or meets local standards for surgical repair or interventional dilation.
   3. A history of prior renal artery intervention including balloon angioplasty or stenting.
   4. Multiple main renal arteries in either kidney.
2. Individual has an estimated glomerular filtration rate (eGFR) of < 30mL/min/1.73m2, using the MDRD calculation.
3. Individual has type 1 diabetes mellitus.
4. Individual has experienced a myocardial infarction, or a cerebrovascular accident within 6 months of the screening visit, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
5. Individual has a scheduled or planned surgery or cardiovascular intervention in the next 6 months.
6. Individual has hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous.
7. Individual has an implantable cardioverter defibrillator (ICD) or pacemaker, or any other metallic implant which is not compatible with magnetic resonance imaging (MRI).
8. Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia, or arrhythmias such as atrial fibrillation).
9. Individual is pregnant, nursing or planning to be pregnant. [Female participants of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to treatment.]
10. Individual is currently enrolled in another investigational drug or device trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2017-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chieh Suai Tan, M.B.B.S, Principal Investigator — Singapore General Hospital; Soo Teik Lim, M.B.B.S, Principal Investigator — National Heart Centre of Singapore
Locations (2):
- Singapore (2):
  - National Heart Centre of Singapore, Singapore
  - Singapore General Hospital, Singapore